CLINICAL TRIAL: NCT06612541
Title: Point-of-Care Ophthalmic Diagnostic Imaging of Retinopathy of Prematurity
Acronym: ROP Imaging
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Irina De la Huerta, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 231251
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Retinopathy of Prematurity (ROP); ROP Examination
Keywords: Retinopathy of Prematurity; ROP; Prematurity; OCT Imaging
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this proposal is to develop novel HH-SECTR technology for visualizing and quantifying diagnostic disease features in prematurely born infant retinopathy of prematurity (ROP) patients that lead to more informed clinical decision making. Providing depth-resolved vascular information has not been adequately investigated for its diagnostic potential. Furthermore, we seek to identify disease features not currently accessible by standard examination methods to better inform clinical decisions.

DETAILED DESCRIPTION:
Imaging studies using HH-SECTR will be performed to assess and quantify structural and vascular disease features associated with ROP. Weekly HH-SECTR imaging will be performed concurrently with standard-of-care weekly ROP screening. No additional treatments will be given to study patients to benefit HH-SECTR imaging (e.g., sedation, dilation, etc.). Study patients will primarily be imaged in the NICU, but may also be performed under sedation or anesthesia in the operating room concurrent with standard-of-care exams. Because this study will evaluate diagnostic features prognostic of ROP progression and severity, HH-SECTR imaging will be performed until 45 weeks, cessation of ROP screening, or first therapeutic intervention, whichever comes first. Both eyes will undergo HH-SECTR imaging. Diagnostic imaging data will be analyzed following each imaging session. No experimental data will be used to alter the management of patients from the standard-of-care.

Research materials obtained from subjects will include digital HH-SECTR images, digital fundus photography images, and documented examination timeline as part of the standard-of-care. Patient medical records will be used to determine eligibility to participate in the study and will be used as the source documents for following post-examination clinical variables.

The duration of the study will be 5 years. The study records and information will be indefinitely archived per NIH rules using the methods noted above.

ELIGIBILITY:
Inclusion Criteria:

* Preterm male and female infants born at 24-34 weeks gestational age and weighing <1500g at birth

Exclusion Criteria:

* Infants surgically treated for ROP
* Infants with significant health concern that would preclude noninvasive retinal imaging as noted by the primary inpatient team

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm male and female infants born at 24-34 weeks gestational age and weighing <1500g at birth.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Retinal imaging in pediatric ROP patients | Weekly imaging until 45 weeks, cessation of ROP screening, or first therapeutic intervention, whichever comes first
  Real-time noninvasive optical imaging of the retina will be performed out to the ora serrata and ROP diagnostic markers will be evaluated in post-processing and compared against clinical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States